CLINICAL TRIAL: NCT03798535
Title: First Real-world Data on Unresectable Stage III NSCLC Patients Treated With Durvalumab After Chemoradiotherapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4194R00005
Record Dates: First submitted 2018-12-21; First posted 2019-01-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This is a non-interventional/observational cohort of unresectable Stage III NSCLC patients treated with durvalumab.

The study will be carried out as a retrospective review of established medical records of unresectable Stage III NSCLC patients treated with durvalumab.

DETAILED DESCRIPTION:
This is a non-interventional/observational study including unresectable Stage III NSCLC patients treated with durvalumab. Patients will be selected from the following participating countries: Australia, Belgium, Israel, Netherlands, Norway, France, Germany, Italy, Switzerland, Spain* and the United Kingdom.

Chart abstractions will occur at specified intervals up to five years after the patient had the first dose of durvalumab. A target of four (maximum five) chart extractions is anticipated for each participant. Dates may be adjusted based on local market ethics processes or patient enrolment.

* First chart extraction will be used to determine which patients meet the inclusion/exclusion criteria for the study and will retrospectively collect all data from diagnosis of unresectable Stage III NSCLC to durvalumab start date (index date).
* The second chart extraction will be triggered at time of estimated maturity of PFS data.
* The third chart extraction will be triggered at time of estimated maturity of OS data.
* The fourth (final) chart extractions will occur 5-years after EAP enrolment to provide final PFS and OS data, together with updated results for all secondary and descriptive endpoints.
* The dates for the second through fourth chart abstractions may be adjusted, pending data availability. The estimated PFS and OS maturity will be calculated from the actual patient index dates (date of first dose of durvalumab) together with the distribution of PFS and OS observed in the PACIFIC trial.

  * Spain only contributed to DE1 and DE2.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or any locally required authorisation obtained from the patient prior to performing any protocol-related procedures
* Age ≥ 18 years at time of study entry or adult according to each country regulations for age of majority
* Patients must have histologically or cytologically documented diagnosis of NSCLC with a locally advanced, or locally recurrent, unresectable (stage III) disease (according to American Joint Committee on Cancer [AJCC] lung cancer edition 7 or 8)
* Patients must have been enrolled in one of the durvalumab EAPs Patients must have been treated with at least one dose of durvalumab within the EAP prior to the study entry and between start of EAP in the country, from September 2017 or later up to end of EAP enrolment or MA + three months (estimated as maximum to 30 December 2018) (whichever occurs earlier).

Patients who die during the EAP are eligible to enter in the study when local laws allow for a consent waiver, if all other inclusion/exclusion criteria are met.

Exclusion Criteria:

-Patients treated with durvalumab in clinical studies prior to the index date (first dose of durvalumab received within the EAP).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were selected from the following participating countries: Australia, Belgium, Israel, Netherlands, Norway, France, Germany, Italy, Switzerland, Spain* and the United Kingdom. Data will be collected from those patients who have received at least one dose of durvalumab between Sep 2017 through 21 Dec 2018. Patients may participate in other clinical trials during this follow-up period.
  Patients must have completed a platinum-based chemotherapy concurrently or sequentially with radiation therapy without evidence of disease progression. There is no fixed max duration for durvalumab treatment and it continues until the physician determines that it is in the patient's best interest to stop therapy. Later EAP protocol was amended to allow durvalumab treatment duration of no more than 12 months.
  *Spain only contributed to DE1 and DE2.
Sampling Method: Non-Probability Sample
Enrollment: 1156 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Real-world progression free survival (rwPFS) | Patients are followed up from the index date (durvalumab (D) first dose date) to progressive disease (PD), death (if no PD), or loss to follow up if no PD/death. PFS reported at 1, 2, 3, and 5 years after D initiation.
  PFS defined as time from the index date (D first dose date) to the date of investigator-determined disease progression or death (if no progression).
Overall survival (OS) | Patients are followed up from the index date (D first dose date) to death or loss to follow up in the absence of death. OS reported at 2, 3, and 5 years after D initiation.
  OS defined as time from the index date (D first dose date) to the date of death.

SECONDARY OUTCOMES:
Adverse events of special interest | Adverse event data are collected from the time of starting durvalumab (D) throughout the D treatment period up to 90 days after last D infusion or at time of next subsequent therapy initiation (whichever occurred earlier).
  Adverse events of special interest assessed in the study included the following:
  * Diarrhoea / colitis and intestinal perforation
  * Pneumonitis / ILD
  * Hepatitis / transaminase increases
  * Endocrinopathies (i.e., events of hypophysitis / hypopituitarism, adrenal insufficiency, hyper- and hypo-thyroidism and type I diabetes mellitus)
  * Rash / dermatitis
  * Nephritis / blood creatinine increases
  * Pancreatitis / serum lipase and amylase increases
  * Myocarditis
  * Myositis / polymyositis
  * Neuropathy / neuromuscular toxicity (Guillain-Barré, and myasthenia gravis)
  * Other inflammatory responses that are rare / less frequent with a potential immune-mediated aetiology include, but are not limited to, pericarditis, sarcoidosis, uveitis, and other events involving the eye, skin, haematological and rheumatological events.
Time to death or distant metastasis | Patients are followed up from the index date (D first dose date) to distant metastasis (DM), death (if no DM), or loss to follow up if no DM/death. Time to death or DM reported at 1, 2, 3, and 5 years after the D initiation.
  Time to death or DM was defined as time from the index date (D first dose date) to DM or death (if no DM).
Time to death or local recurrence | Patients are followed up from the index date (D first dose date) to local recurrence (LR), death (if no LR), or loss to follow up if no LR/death. Time to death or LR reported at 1, 2, 3, and 5 years after the D initiation.
  Time to death or LR is defined as time from the index date (D first dose date) to LR or death (if no LR).
Time to first subsequent treatment or death | Patients are followed up from the index date (D first dose date) to first subsequent treatment (ST) after D, death (if no ST), or loss to follow up if no ST/death. Time to first ST/death reported at 1, 2, 3, and 5 years after the D initiation.
  Time to first ST or death is defined as time from the index date (D first dose date) to the first ST or death (if no ST).

CONTACTS AND LOCATIONS:
Locations (227):
- Australia (34):
  - Research Site, Ballarat
  - Research Site, Bankstown
  - Research Site, Bedford Park
  - Research Site, Bendigo
  - Research Site, Bentleigh East
  - Research Site, Bowral
  - Research Site, Box Hill
  - Research Site, Campbelltown
  - Research Site, Camperdown
  - Research Site, Canberra
  - Research Site, Clayton
  - Research Site, Coffs Harbour
  - Research Site, Douglas
  - Research Site, Elizabeth Vale
  - Research Site, Frankston
  - Research Site, Hamlyn Terrace
  - Research Site, Hervey Bay
  - Research Site, Hobart
  - Research Site, Joondalup
  - Research Site, Kingswood
  - Research Site, Liverpool
  - Research Site, Malvern
  - Research Site, Melbourne
  - Research Site, Murdoch
  - Research Site, Orange
  - Research Site, Rockhampton
  - Research Site, St Leonards
  - Research Site, Subiaco
  - Research Site, Traralgon
  - Research Site, Tugun
  - Research Site, Warrnambool
  - Research Site, Wendouree
  - Research Site, Westmead
  - Research Site, Wollongong
- Belgium (21):
  - Research Site, Aalst
  - Research Site, Bouge
  - Research Site, Braine-l'Alleud
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Dendermonde
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Herstal
  - Research Site, Heusden-Zolder
  - Research Site, Ieper
  - Research Site, Kuringen
  - Research Site, Liège
  - Research Site, Loverval
  - Research Site, Mons
  - Research Site, Ottignies
  - Research Site, Roeselare
  - Research Site, Ronse
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Truiden
  - Research Site, Yvoir
- France (57):
  - Research Site, Abbeville
  - Research Site, Aix-en-Provence
  - Research Site, Albi
  - Research Site, Antony
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Brest
  - Research Site, Carcassonne
  - Research Site, Chauny
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Contamine-sur-Arve
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Gap
  - Research Site, Grenoble
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, Le Mans
  - Research Site, Levallois-Perret
  - Research Site, Libourne
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lorient
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Mâcon
  - Research Site, Metz-Tessy
  - Research Site, Montpellier
  - Research Site, Morlaix
  - Research Site, Muret
  - Research Site, Nancy
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Périgueux
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Tarbes
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Valence
  - Research Site, Vantoux
  - Research Site, Villefranche-sur-Saône
- Germany (24):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bremen
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Fürth
  - Research Site, Georgsmarienhütte
  - Research Site, Gütersloh
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Immenhausen
  - Research Site, Kaiserslautern
  - Research Site, Karlsruhe
  - Research Site, Kempten
  - Research Site, München
  - Research Site, Münnerstadt
  - Research Site, Oldenburg
  - Research Site, Paderborn
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Würselen
- Israel (11):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Nazareth
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (42):
  - Research Site, Alessandria
  - Research Site, Ancona
  - Research Site, Arezzo
  - Research Site, Aviano
  - Research Site, Bari
  - Research Site, Bolzano
  - Research Site, Brescia
  - Research Site, Catanzaro
  - Research Site, Feltre
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Imola
  - Research Site, La Spezia
  - Research Site, Lecce
  - Research Site, Lido di Camaiore
  - Research Site, L’Aquila
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Mirano
  - Research Site, Modena
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Pistoia
  - Research Site, Ravenna
  - Research Site, Reggio Emilia
  - Research Site, Rimini
  - Research Site, Rionero in Vulture
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Sora
  - Research Site, Terni
  - Research Site, Treviglio
  - Research Site, Trieste
  - Research Site, Udine
  - Research Site, Varese
  - Research Site, Verona
- Netherlands (19):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Heerlen
  - Research Site, Hilversum
  - Research Site, Leiden
  - Research Site, Maastricht
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, The Hague
  - Research Site, Utrecht
  - Research Site, Zutphen
- Norway (4):
  - Research Site, Arendal
  - Research Site, Drammen
  - Research Site, Oslo
  - Research Site, Tromsø
- Switzerland (7):
  - Research Site, Altdorf
  - Research Site, Bülach
  - Research Site, Chur
  - Research Site, Fribourg
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Neuchâtel
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Colchester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Poole
  - Research Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Langberg CW, Horndalsveen H, Helland A, Haakensen VD. Factors associated with failure to start consolidation durvalumab after definitive chemoradiation for locally advanced NSCLC. Front Oncol. 2023 Jul 5;13:1217424. doi: 10.3389/fonc.2023.1217424. eCollection 2023. PMID 37476372
- [Derived] Zhao B, Li H, Ma W. Durvalumab After Chemoradiotherapy for Patients With Unresectable Stage III NSCLC: The PACIFIC-R Study. J Thorac Oncol. 2023 Apr;18(4):e38-e39. doi: 10.1016/j.jtho.2022.11.002. No abstract available. PMID 36990576
- [Derived] Girard N, Bar J, Garrido P, Garassino MC, McDonald F, Mornex F, Filippi AR, Smit HJM, Peters S, Field JK, Christoph DC, Sibille A, Fietkau R, Haakensen VD, Chouaid C, Markman B, Hiltermann TJN, Taus A, Sawyer W, Allen A, Chander P, Licour M, Solomon B. Treatment Characteristics and Real-World Progression-Free Survival in Patients With Unresectable Stage III NSCLC Who Received Durvalumab After Chemoradiotherapy: Findings From the PACIFIC-R Study. J Thorac Oncol. 2023 Feb;18(2):181-193. doi: 10.1016/j.jtho.2022.10.003. Epub 2022 Oct 25. PMID 36307040
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194R00005&attachmentIdentifier=54f53e57-7310-4d49-ac77-d5057aa4f7ca&fileName=D4194R00005_PACIFICR_CSR_Synopsis_redacted.pdf&versionIdentifier=